CLINICAL TRIAL: NCT02174822
Title: A Phase 1, Single-center, Open-label, Sequential Drug Interaction Study Between AVP-786 (Deuterated [d6] Dextromethorphan Hydrobromide [DM]/Quinidine Sulfate [Q]) and Paroxetine and Between AVP-786 and Duloxetine in Healthy Subjects
Brief Title: A Phase 1, Drug Interaction Study Between AVP-786 and Paroxetine and Between AVP-786 and Duloxetine in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 14-AVP-786-101
Record Dates: First submitted 2014-06-23; First posted 2014-06-26 (Estimated); Last update posted 2022-02-18 (Actual); Status verified 2014-06

CONDITIONS: Drug-drug Interaction
Keywords: Drug-drug interaction; Pharmacokinetics; Healthy Volunteers; deuterated dextromethorphan; deuterated dextromethorphan with quinidine
MeSH Terms: interventions — Paroxetine; Duloxetine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Paroxetine + AVP-786 (Experimental): Paroxetine once daily orally Days 1-20. AVP-786 twice daily orally for Days 13 - 20.
  Interventions: Drug: AVP-786; Drug: Paroxetine
- AVP-786 + paroxetine (Experimental): AVP-786 twice daily orally Days 1-20. Paroxetine once daily orally for Days 9 - 20
  Interventions: Drug: AVP-786; Drug: Paroxetine
- Duloxetine + AVP-786 (Experimental): Duloxetine twice daily orally Days 1 - 13. AVP-786 twice daily orally Days 6 - 13.
  Interventions: Drug: AVP-786; Drug: Duloxetine
- AVP-786 + duloxetine (Experimental): AVP-786 twice daily orally Days 1 - 13. Duloxetine twice daily Days 9 - 13.
  Interventions: Drug: AVP-786; Drug: Duloxetine

INTERVENTIONS:
Drug: AVP-786
Drug: Paroxetine
  Arms: AVP-786 + paroxetine; Paroxetine + AVP-786
Drug: Duloxetine
  Arms: AVP-786 + duloxetine; Duloxetine + AVP-786

SUMMARY:
To assess steady state pharmacokinetics (PK), safety and tolerability between AVP-786 (deuterated [d6] dextromethorphan hydrobromide [DM]/quinidine sulfate [Q]) and paroxetine and between AVP-786 and duloxetine.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult males and females
* 18 - 50 years of age
* BMI 18 - 30 kg/m2

Exclusion Criteria:

* History or presence of significant disease
* History of substance abuse and/or alcohol abuse with the past 3 years
* Use of tobacco-containing or nicotine-containing products within 6 months
* Use of any prescription or the over-the-counter medications within 14 days

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2014-01; Primary Completion 2014-03 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Change in plasma concentrations of paroxetine after combined dosing with AVP-786 paroxetine in healthy subjects | 20 days
Change in plasma concentration of AVP-786 (parent and metabolites) after dosing in combination with paroxetine. | 20 days
Change in plasma concentration of duloxetine after combined dosing with AVP-786 | 13 days
Change in plasma concentration of AVP-786 after combined dosing with duloxetine. | 13 days

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) for AVP-786 and paroxetine | 20 days
Incidence of adverse events (AEs) for AVP-786 and duloxetine | 13 days

CONTACTS AND LOCATIONS:
Overall Officials: Jason Lickliter, MBBS PhD FRACP, Principal Investigator — Nucleus Network
Locations (1):
- Nucleus Network, Melbourne, Victoria, Australia